CLINICAL TRIAL: NCT04926935
Title: Bloodstram Infections in Intensive Care Unit. A Single Centre Bacteriological Analysis Between 2007-2019.
Brief Title: Bloodstram Infections in ICU. Single Centre Observational Study.
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, Associate Professor, Military Institute od Medicine National Research Institute
Other Study IDs: 09
Record Dates: First submitted 2021-06-04; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Bloodstream Infection; Antibiotic Resistant Strain; Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized in the ICU during the study period.: Patients hospitalized in the ICU during the study period with clinically suspected infection.
  Interventions: Diagnostic Test: Microbiological analysis of blood samples.

INTERVENTIONS:
Diagnostic Test: Microbiological analysis of blood samples. — Microbiological analysis of blood samples collected from the patients with clinically suspected infection.

SUMMARY:
Hospital-acquired bloodstream infection (BSI) is serious care problem worldwide associated with significant morbidity and mortality. However, only few nationwide studies have focused on the incidence of BSI, and its results were often inconsistent.

The objective of this study was to analyze bloodstream infections in patients hospitalized in the intensive care unit of the tertiary, university hospital. Special attention was put on the etiology of the infections, the antimicrobial susceptibility/resistance of the isolated pathogens, as well as the incidence of central vein catheters infections in the analyzed population.

Data were collected in the intensive care unit of the Military Institute of Medicine, Warsaw, Poland, between January, 1, 2007 and December, 31, 2019.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in the ICU with clinically suspected infection.

Exclusion Criteria:

* none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in the ICU with clinically suspected infection between 2007-2019.
Sampling Method: Probability Sample
Enrollment: 3502 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Results of microbiological analysis. | After completion of the microbiological analysis, up to 72 hours.
  Results of the microbiological analysis of the blood samples collected from patients with clinically suspected infections hospitalized in the ICU during the study period.
Isolated pathogens' susceptibility for antimicrobial agents. . | After completion of the microbiological analysis, up to 72 hours.
  Results of the microbiological analysis of the blood samples collected from patients with clinically suspected infections hospitalized in the ICU during the study period.
Isolated pathogens' resistance for antimicrobial agents. . | After completion of the microbiological analysis, up to 72 hours.
  Results of the microbiological analysis of the blood samples collected from patients with clinically suspected infections hospitalized in the ICU during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Tomaszewski, MD, PhD, Principal Investigator — Military Institute od Medicine National Research Institute
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garrouste-Orgeas M, Timsit JF, Tafflet M, Misset B, Zahar JR, Soufir L, Lazard T, Jamali S, Mourvillier B, Cohen Y, De Lassence A, Azoulay E, Cheval C, Descorps-Declere A, Adrie C, Costa de Beauregard MA, Carlet J; OUTCOMEREA Study Group. Excess risk of death from intensive care unit-acquired nosocomial bloodstream infections: a reappraisal. Clin Infect Dis. 2006 Apr 15;42(8):1118-26. doi: 10.1086/500318. Epub 2006 Mar 14. PMID 16575729
- [Result] Laupland KB, Lee H, Gregson DB, Manns BJ. Cost of intensive care unit-acquired bloodstream infections. J Hosp Infect. 2006 Jun;63(2):124-32. doi: 10.1016/j.jhin.2005.12.016. Epub 2006 Apr 18. PMID 16621137
- [Result] Wilson J, Elgohari S, Livermore DM, Cookson B, Johnson A, Lamagni T, Chronias A, Sheridan E. Trends among pathogens reported as causing bacteraemia in England, 2004-2008. Clin Microbiol Infect. 2011 Mar;17(3):451-8. doi: 10.1111/j.1469-0691.2010.03262.x. PMID 20491834
- [Result] Nielsen SL, Pedersen C, Jensen TG, Gradel KO, Kolmos HJ, Lassen AT. Decreasing incidence rates of bacteremia: a 9-year population-based study. J Infect. 2014 Jul;69(1):51-9. doi: 10.1016/j.jinf.2014.01.014. Epub 2014 Feb 25. PMID 24576825
- [Result] de Kraker ME, Jarlier V, Monen JC, Heuer OE, van de Sande N, Grundmann H. The changing epidemiology of bacteraemias in Europe: trends from the European Antimicrobial Resistance Surveillance System. Clin Microbiol Infect. 2013 Sep;19(9):860-8. doi: 10.1111/1469-0691.12028. Epub 2012 Oct 8. PMID 23039210
- [Result] Goto M, Al-Hasan MN. Overall burden of bloodstream infection and nosocomial bloodstream infection in North America and Europe. Clin Microbiol Infect. 2013 Jun;19(6):501-9. doi: 10.1111/1469-0691.12195. Epub 2013 Mar 8. PMID 23473333